CLINICAL TRIAL: NCT00951613
Title: A Phase II Study of NK012 in Sensitive Relapsed and Refractory Relapsed Small-Cell Lung Cancer (SCLC)
Brief Title: A Study of NK012 in Patients With Relapsed Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nippon Kayaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6012212US
Record Dates: First submitted 2009-05-21; First posted 2009-08-04 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell lung cancer; carcinoma, lung; Sensitive-relapsed or refractory-relapsed small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: NK012 — 30 minute IV infusion once every 28 days. NK012 dose is 28 mg/m^2 (or 18 mg/m^2 depending on UGT1A1 polymorphism, with potential to dose escalate). Dose escalation cannot exceed 28 mg/m^2. Dosing will proceed until progression or unacceptable toxicity develops, or decision by patient or investigator to stop.

SUMMARY:
The purpose of this study is to determine whether NK012 is safe and effective in the treatment of relapsed small cell lung cancer.

DETAILED DESCRIPTION:
This is a Phase II, open label, single arm, multicenter study of NK012 in patients with sensitive relapsed SCLC (at least 90 days since first line therapy) or refractory relapsed SCLC (< 90 days since first line therapy). NK012 will be administered by intravenous infusion over 30 minutes once every 28 days (on Day 1 of each cycle). Patients will be screened for UGT1A1 polymorphism prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of SCLC, which has relapsed after first line chemotherapy for extensive-stage SCLC or first-line chemoradiotherapy for limited-stage SCLC.
2. Have received one, and only one, prior chemotherapy or chemoradiotherapy regimen for either newly diagnosed extensive-stage disease or limited-stage disease.
3. Prior therapies must be completed at least 4 weeks prior to enrollment and patients must have recovered from all acute toxicities.
4. Measurable disease by RECIST.
5. ECOG performance status of 0-2.
6. At least 18 years of age.
7. Adequate bone marrow function as defined by absolute neutrophil count of greater than or equal to 1,500/mm^3 and platelets of greater than or equal to 100,000/mm^3.
8. AST (SGOT) and ALT (SGPT) levels no greater than 3 x the institutional ULN, and total bilirubin less than or equal to 1.5 x ULN.
9. Serum creatinine less than or equal to 1.5 x ULN, or creatinine clearance greater than or equal to 60 mL/min (Cockcroft-Gault formula) for patients with serum creatinine levels > 1.5 x ULN.
10. Able to understand and show willingness to sign a written informed consent document.

Exclusion criteria:

1. Patient has Gilbert's Syndrome.
2. Prior chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
3. Lack of recovery from adverse effects due to agents administered more than 4 weeks prior to study entry.
4. Concurrent use of other investigational agent.
5. History of brain metastases or spinal cord compression, unless irradiated a minimum of 4 weeks before study entry and stable without requirement for corticosteroids for > 1 week.
6. Prior exposure to topoisomerase 1 inhibitors (i.e., irinotecan, topotecan, camptothecin).
7. Concurrent serious infections requiring parenteral therapy.
8. Pregnant or of childbearing potential and not using methods to avoid pregnancy. A negative pregnancy test (urine or serum) must be documented at baseline for women of childbearing potential. Patients may not breast-feed infants while on this study.
9. Significant cardiac disease including heart failure that meets New York Heart Association (NYHA) class III and IV definitions, history of myocardial infarction within one year of study entry, uncontrolled dysrhythmias or poorly controlled angina.
10. History of serious ventricular arrhythmia (VT or VF, greater than or equal to 3 beats in a row), QTc greater than or equal to 450 msec for men and 470 msec for women, or LVEF less than or equal to 40% by MUGA or ECHO.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-07; Primary Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the overall antitumor activity (overall response rate) of NK012 | At baseline and after every 2 cycles; PR or CR must be confirmed no less than 4 weeks after the first response was recorded

SECONDARY OUTCOMES:
Progression-free survival | Monthly for 6 months after patient goes off study, then every 3 months thereafter
Duration of response | Monthly for 6 months after patient goes off study, then every 3 months thereafter
Overall survival | Monthly for 6 months after patient goes off study, then every 3 months thereafter
Toxicity profile of NK012 | Duration of study and up to 30 days after off-study

CONTACTS AND LOCATIONS:
Overall Officials: David R Spigel, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Sarah Cannon Research Institute, Nashville, Tennessee, United States